CLINICAL TRIAL: NCT06422403
Title: A Value-Driven Study on Reducing Immune Checkpoint Inhibitor Dosing Frequency in Advanced Cancers: Phase 2 Randomized Trial (VALUE-CHECK)
Brief Title: A Value-Driven Study on Reducing Immune Checkpoint Inhibitor Dosing Frequency in Advanced Cancers
Acronym: VALUE-CHECK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-3881
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Hepatocellular; Gastric Adenocarcinoma; GastroEsophageal Cancer; Oesophageal Cancer; Non-small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: Nivolumab; Atezolizumab; Pembrolizumab; Extended dosing interval
MeSH Terms: conditions — Carcinoma, Hepatocellular; Esophageal Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: This study is a prospective, open label, multi-centre phase 2 trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort A (SOC) (Active Comparator): Nivolumab, XELOX/FOLFOX
  Interventions: Drug: Standard of Care - A
- Cohort A (EDI) (Experimental): Nivolumab, XELOX/FOLFOX
  Interventions: Drug: Extended Dosing Interval - A
- Cohort B (SOC) (Active Comparator): Bevacizumab, Atezolizumab
  Interventions: Drug: Standard of Care - B
- Cohort B (EDI) (Experimental): Bevacizumab, Atezolizumab
  Interventions: Drug: Extended Dosing Interval - B
- Cohort C (SOC) (Active Comparator): Pembrolizumab
  Interventions: Drug: Standard of Care - C
- Cohort C (EDI) (Experimental): Pembrolizumab
  Interventions: Drug: Extended Dosing Interval - C

INTERVENTIONS:
Drug: Extended Dosing Interval - A — Nivolumab 360mg 6 weekly (up to 2 years) + XELOX Nivolumab 240mg 4 weekly (up to 2 years) + FOLFOX
  Arms: Cohort A (EDI)
Drug: Extended Dosing Interval - B — Bevacizumab + Atezolizumab 1200mg 6 weekly (up to 2 years)
  Arms: Cohort B (EDI)
Drug: Extended Dosing Interval - C — Pembrolizumab 200mg 6 weekly (up to 2 years)
  Arms: Cohort C (EDI)
Drug: Standard of Care - A — Nivolumab 360mg 3 weekly (up to 2 years) + XELOX Nivolumab 240mg 2 weekly (up to 2 years) + FOLFOX
  Arms: Cohort A (SOC)
Drug: Standard of Care - B — Bevacizumab + Atezolizumab 1200mg 3 weekly (up to 2 years)
  Arms: Cohort B (SOC)
Drug: Standard of Care - C — Pembrolizumab 200mg 3 weekly (up to 2 years)
  Arms: Cohort C (SOC)

SUMMARY:
This study is a prospective, open label, multi-centre phase 2 trial which assesses the efficacy and safety of standard dosing compared to extended dosing interval of nivolumab, atezolizumab or pembrolizumab in advanced/unresectable gastric/gastroesophageal junction/oesphageal adenocarcinomas with PDL1 CPS ≥5%, hepatocellular carcinoma andnon-small cell lung cancer with PDL1 TPS≥50% with no prior treatment. The investigators hypothesize that nivolumab, pembrolizumab and atezolizumab can be used efficiently at extended dosing intervals, compared to their approved labels with comparable clinical outcome.

DETAILED DESCRIPTION:
This study aims to assess the noninferiority of progression free survival of standard dosing compared to extended dosing interval of nivolumab, pembrolizumab and atezolizumab in advanced/unresectable gastric/gastroesophageal junction/oesphageal adenocarcinomas with PDL1 CPS ≥5%, hepatocellular carcinoma, and non-small cell lung cancer with PDL1 TPS≥50%.

Secondary Objective

* To investigate the safety, overall survival (OS) of ICI at extended dosing interval of the standard versus extended dosing interval groups.
* To investigate the pharmacokinetics (PK) of nivolumab, atezolizumab or pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study-specific procedure
2. Patients with one of the following:

   * Cohort A: Previously untreated locally advanced/metastatic HER2 -ve gastric/gastroesophageal junction/esophageal (PDL1 CPS ≥5% adenocarcinomas not amenable to curative surgery or radiotherapy who are above to begin platinum double and nivolumab.
   * Cohort B: Previously untreated locally advanced/metastatic Child's A hepatocellular carcinoma not amenable to curative surgery or radiotherapy who are above to begin atezolizumab and bevacizumab.
   * Cohort C: Previously untreated locally advanced/metastatic lung adenocarcinoma (PDL1 TPS≥50%, EGFR/ALK wildtype) not amenable to curative surgery or radiotherapy who are above to begin pembrolizumab monotherapy
3. Measurable disease per RECIST 1.1 criteria
4. ECOG Performance status is 0-2
5. Normal organ and bone marrow function measured within 28 days before the study as defined below:

   * Haemoglobin ≥ 8.0 g/dL and no blood transfusions in the 28 days prior to entry
   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   * No features suggestive of MDS/AML on peripheral blood smear
   * White blood cells (WBC) > 3x10^9/L
   * Platelet count ≥ 100 x 10^9/L
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
   * Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN)
6. A life expectancy ≥ 12 weeks in all patients.
7. Females in childbearing age should be using adequate contraceptive measures, should not be breastfeeding and their pregnancy test prior to the start of treatment must be negative. Evidence of non-child-bearing potential is fulfilled by one of the following criteria at screening:
8. The post-menopausal period defined as age ≥50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
9. Women <50 years old they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range.
10. Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not a tubal ligatio
11. Male patients should be willing to use barrier contraception
12. The patient is willing to comply with the protocol during the study including undergoing treatment and scheduled visits and examinations including follow up.
13. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and is considered suitable for accurate repeated measurements

Exclusion Criteria:

1. Patients who have previously received immune checkpoint inhibitors or investigational monoclonal antibody therapy.
2. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years
3. Unstable spinal cord compression/brain metastases unless asymptomatic and not requiring steroids for at least 2 weeks prior to the start of study treatment. For patients with brain metastases, gamma knife or stereotactic brain surgery is allowed prior to study treatment.
4. Major surgery within 4 weeks of starting study treatment and patients must have recovered from any effects of any major surgery. Minor surgery is allowed.
5. Severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which based on investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or having active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
6. Autoimmune disorders
7. Males and females of reproductive potential who are not using an effective method of contraception and females who are pregnant or breastfeeding or have a positive serum pregnancy test prior to study entry
8. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
9. Previous allogeneic bone marrow transplant.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from date of first dosing until the date of objective disease progression as defined by Response Evaluation Criteria in Solid Tumor (RECIST 1.1) or death (by any cause in the absence of progression).

SECONDARY OUTCOMES:
Number of participant with treatment related haematological and non-haematological toxicities | Up to 2 years
  As defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Objective response rate | Up to 2 years
  Percentage of patients who have at least one confirmed response of 'complete response' or 'partial response' as defined by Response Evaluation Criteria in Solid Tumor (RECIST 1.1), that is confirmed at least 4 weeks later
Duration of Response | Up to 2 years
  Duration of response will be defined as the time from the date of first documented response, that is subsequently confirmed until the date of documented progression or death in the absence of disease progression, the end of response should coincide with the date of progression or death from any cause used for the PFS endpoint.
Disease control rate | Up to 2 years
  Disease control rate is defined as the proportion of patients with a best overall response of CR = complete response, PR = partial response, or SD = stable disease, as defined by Response Evaluation Criteria in Solid Tumor (RECIST 1.1)
Overall survival | Up to 2 years
  Overall survival will be assessed based on the date of first dose and survival status at the time of analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Department of Hematology-Oncology, National University Hospita, Singapore, Singapore